CLINICAL TRIAL: NCT00647036
Title: Microbial Invasion During Parenteral Nutrition in Surgical Infants Receiving Glutamine.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Institute of Child Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Other
Other Study IDs: 07SG10
Record Dates: First submitted 2008-03-26; First posted 2008-03-31 (Estimated); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Surgical Infants Requiring Total Parenteral Nutrition
Keywords: Parenteral nutrition, Infants, Dipeotiven, Microbial invasion
MeSH Terms: conditions — Hyperphagia | interventions — alanylglutamine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Dipeptiven (L-glutamine- Lalanine)
  Interventions: Drug: Dipeptiven (L-glutamine- Lalanine)
- 2 (Placebo Comparator): Isonitrogenous Vaminolact
  Interventions: Dietary Supplement: Isonitrogenous Vaminolact

INTERVENTIONS:
Dietary Supplement: Isonitrogenous Vaminolact — Isonitrogenous Vaminolact
  Arms: 2
Drug: Dipeptiven (L-glutamine- Lalanine) — 0.6g/kg/day
  Arms: 1

SUMMARY:
We hypothesise that the addition of glutamine supplementation to both parenteral nutrition and enteral feeds in surgical newborn infants leads to a reduction in bacterial invasion.

ELIGIBILITY:
Inclusion Criteria:

* Infants who have undergone surgical procedures for congenital anomalies or
* Intestinal inflammation who require total parenteral nutrition.

Exclusion Criteria:

-

Max Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2009-07 (Actual); Primary Completion 2011-12 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Evidence of microbial invasion | 5 days

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Child Health, 30 Guilford Street, London, United Kingdom

REFERENCES:
- [Result] Bishay M, Simchowitz V, Harris K, Macdonald S, De Coppi P, Klein N, Eaton S, Pierro A; MIGS Trial Group. The Effect of Glutamine Supplementation on Microbial Invasion in Surgical Infants Requiring Parenteral Nutrition: Results of a Randomized Controlled Trial. JPEN J Parenter Enteral Nutr. 2020 Jan;44(1):80-91. doi: 10.1002/jpen.1700. Epub 2019 Sep 9. PMID 31502272